CLINICAL TRIAL: NCT02147925
Title: Efficacy of Liraglutide vs. Sitagliptin vs. Insulin Glargine Per Day on Liver Fat When Combined With Metformin in T2DM Subjects With Non-alcoholic Fatty-liver Disease
Brief Title: Efficacy Study of Liraglutide vs.Sitagliptin vs. Glargine on Liver Fat in T2DM Subjects
Acronym: LIGHT-ON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianping Weng, professor, vice president, the third affiliated hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS201404
Record Dates: First submitted 2014-05-16; First posted 2014-05-28 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2017-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; Glucagon-like peptide-1 receptor agonists; Diabetes mellitus, type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Metformin; Liraglutide; Insulin Glargine; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liraglutide (Active Comparator): Liraglutide combined with metformin
  Interventions: Drug: Liraglutide combined with metformin
- Insulin glargine (Active Comparator): Insulin glargine combined with metformin
  Interventions: Drug: Insulin glargine combined with metformin
- Sitagliptin (Active Comparator): Sitagliptin combined with metformin
  Interventions: Drug: Sitagliptin combined with metformin

INTERVENTIONS:
Drug: Liraglutide combined with metformin — Liraglutide, 0.6mg per day for the first week, and will be increased to 1.2mg per day for the second week, and finally 1.8mg per day since the third week
  Other Names: Victoza®, Novo Nordisk
  Arms: Liraglutide
Drug: Insulin glargine combined with metformin — The initial dose will be 0.2 unit/kg/d
  Other Names: Lantus®, Sanofi
  Arms: Insulin glargine
Drug: Sitagliptin combined with metformin — The dose throughout the study will be 100mg per day.
  Other Names: Januvia®, Merck & Co. Inc.
  Arms: Sitagliptin

SUMMARY:
The aim of this study is to explore the effectiveness of liraglutide combined with metformin in non-alcoholic fatty-liver disease patients with type 2 diabetes mellitus (T2DM) compared to sitagliptin and insulin glargine in combination with metformin.

DETAILED DESCRIPTION:
This is a 26-week, randomized, open-label, active controlled, parallel group, multi-centre trial.To compare the change of intrahepatic lipids (IHL) as measured by magnetic resonance spectroscopy(MRS) or MRI estimated proton density fat fraction (MRI-PDFF) as measured by MRI IDEAL IQ (Iterative Decomposition of water andfat with Echo Asymmetryand Least-squares estimation) in type 2 diabetic patients with non-alcoholic fatty-liver disease after a 26-week treatment of liraglutide, sitagliptin or insulin glargine per day combined with metformin.The primary endpoint will be defined by intrahepatic lipids (IHL) as measured by magnetic resonance spectroscopy (MRS) or MRI-PDFF as measured by MRI IDEAL IQ.

ELIGIBILITY:
Inclusion Criteria:

* Recorded Type 2 diabetes diagnosed at least 3 months before the study; At least 3 months treatment on a stable dose（≧1500mg/d）of metformin before the study
* 6.5%<HbA1c ≤10%
* Clinically diagnosed simple liver steatosis
* 30-75 years old
* Female subjects should be postmenopausal, surgically sterile, or using contraceptives for 3 months before screening and continuing throughout the study;
* BMI 20~35 kg/m2 and with a history of stable body weight (≤10%variation for ≥3 months)
* intrahepatic lipids (IHL) >10%

Exclusion Criteria:

* Type 1 diabetes
* Treatment within the last 3 months with Thiazolidinediones(TZDs), orlistat, insulin, any history of incretin based therapy or any other drugs associated with hepatic steatosis (including but not limited to glucocorticoids, tamoxifen, amiodarone or methotrexate)
* History or current episode of pancreatitis or other disease of the pancrea; Impaired liver function, defined as plasma alanine transaminase(ALT) >2.5 times of upper normal limit
* Moderate and severe renal insufficiency defined as MDRD formula glomerular filtration rate<60ml/min/1.73m2
* Weekly alcohol intake>14 units for women or >21 units for men
* Any history of liver disease including metabolic or auto-immune liver diseases or viral hepatitis
* History or family history of medullary thyroid cancer(MTC), or multiple endocrine neoplasia type 2(MEN-2)
* Congestive heart failure(NYHA III~IV)
* Severe gastric-intestinal diseases
* Pregnancy and/or intention of becoming pregnant
* Known proliferative retinopathy or maculopathy requiring acute treatment as judged by the Investigator; Use of non-herbal Chinese medicine or other non-herbal local medicine with unknown/unspecified content. Herbal traditional Chinese medicine or other local herbal medicines may, at the Investigator's discretion, be continued throughout the trial at an unchanged dose

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Intrahepatic lipids (IHL) | 26-week
  To compare the change of intrahepatic lipids (IHL) in type 2 diabetic patients with non-alcoholic fatty-liver disease after a 26-week treatment of liraglutide, sitagliptin or insulin glargine per day combined with metformin.

SECONDARY OUTCOMES:
Change of abdominal subcutaneous adipose tissue(SAT) | 26 weeks
  To compare the change of SAT in type 2 diabetic patients
Change of visceral adipose tissue(VAT) | 26 weeks
  To compare the change of VAT in type 2 diabetic patients
Change in hemoglobin A1c(HbA1c) | 26 weeks
  To compare the change of HbA1c in type 2 diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Weng, Doctor, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China